CLINICAL TRIAL: NCT01656187
Title: Attenuation of Corticosteroid Induced Hippocampal Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 032011-007; 1R01DA029596 (NIH)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Organic Memory Impairment
Keywords: memantine; cognition; corticosteroid; prednisone; memory; hippocampus
MeSH Terms: interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine, Then Placebo (Experimental): Participants first received Memantine 10 mg capsule twice a day for 24 weeks. After a washout period of 4 weeks, they then received Placebo capsule (matching Memantine 10 mg capsule) twice a day for 24 weeks.
  Interventions: Drug: Memantine 10 mg capsule; Drug: Memantine-matched Placebo capsule
- Placebo, Then Memantine (Experimental): Participants first received Placebo capsule (matching Memantine 10 mg capsule) twice a day for 24 weeks. After a washout period of 4 weeks, they then received Memantine 10 mg capsule twice a day for 24 weeks.
  Interventions: Drug: Memantine 10 mg capsule; Drug: Memantine-matched Placebo capsule

INTERVENTIONS:
Drug: Memantine 10 mg capsule — Memantine oral capsule was initiated at 5 mg/day at Randomization (Week 0), then titrated to 5 mg twice a day at Week 2, then increased to 10 mg in the morning and 5 mg in the evening at Week 3, and then to 10 mg twice a day (intervention dose) at Weeks 4-24. For the participants in the "Placebo, then Memantine" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
  Other Names: Namenda
Drug: Memantine-matched Placebo capsule — Memantine-matched oral Placebo capsule was initiated at Randomization (Week 0) and maintained Weeks 0-24 in a manner consistent with the active drug titration schedule. The number of placebo capsules matched the number of active drug capsules at each titration checkpoint. For the participants in the "Memantine, then Placebo" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
  Other Names: Sugar pill

SUMMARY:
The purpose of the study is to determine if an investigational drug called memantine,used here as add-on therapy, is associated with improvements in memory, mood and asthma symptoms. We will also examine changes in the brain by taking images or pictures using an MRI/MRS.

DETAILED DESCRIPTION:
A total of 50 outpatients receiving chronic oral corticosteroid therapy will be enrolled in a 52-week randomized, double-blind, placebo-controlled, crossover trial of memantine. Participant will receive either memantine or a placebo for 24 weeks. They have an equal chance of receiving memantine or placebo. After 24 weeks they will discontinue all study medication for 4 weeks. This process will be repeated one additional time in the study and the participant will crossed-over to either memantine or placebo, whichever the participant did not receive before, so they will have taken both placebo and memantine during one of these courses.

Randomization will be stratified by prednisone dose of < 20 mg/day vs. ≥ 20 mg/day. Memantine or placebo starting at 5 milligrams once a day, increased to 5 milligrams twice a day (10 total) at week 2, 15 milligrams total at week 3, and 20 milligrams total from weeks 4-24 unless side effects require the study doctor to increase the initial doses slower than described above or reduce the dose. This same process will be repeated at week 28 after the participant have been completely off of study medication for 4 weeks. Structural MRI and 1HMRS will be obtained at baseline and weeks 24 and 52 (after memantine and placebo).

The clinician version of the structured Clinical Interview for DSM-IV (SCID) is a brief structured interview for major Axis I disorders in DSM-IV including major depressive disorder, dysthymic disorder, bipolar disorders, psychotic disorders, anxiety disorders, eating disorders, and alcohol and substance abuse/dependence. This will be given at baseline to screen for illnesses with CNS involvement or cognitive impairment. Blood draws will be performed at baseline to assess insulin and fasting glucose levels.

Each participant will then return for follow-up appointments as scheduled and repeat outcome measures. Pill counts will be conducted, and a list of current medications and doses will be obtained at each visit. Participants will be evaluated by both the RA and PI at each follow-up appointment.

The HVLT-R will be given at baseline, and weeks 12, 24, 28, 40, and 52; this will be the primary outcome measure. Other cognitive assessments will be performed at these same visits as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any chronic medical condition requiring treatment with oral corticosteroids confirmed by chart review and/or patient assessment by Dr. Khan (co-I).
* Receiving prednisone therapy of at least 5 mg of prednisone/day for at least 6 months with anticipated treatment for ≥ 12 additional months.
* Age 18-65 years.
* Baseline CVLT-II total T score ≤ 54.

Exclusion Criteria:

* Illnesses associated with CNS involvement (e.g., seizures, brain tumors, head injury with loss of consciousness) or cognitive impairment (e.g., substance dependence within the past 2 years, bipolar disorder) Potential participants with mood symptoms secondary to corticosteroids (based on SCID) will not be excluded because this could selectively exclude subjects who are sensitive to the CNS effects of corticosteroids.
* Vulnerable populations (e.g. severe cognitive impairment, pregnant or nursing women, prisoners).
* Severe or life-threatening medical illness that would make completion of study unlikely
* Contraindications to memantine therapy (e.g. severe side effects in the past)
* Danger to self or others as defined by > 1 lifetime suicide attempt or assault, any suicide attempt or assault within the past year, and active suicidal or homicidal ideation with plan and intent.
* Metal implants, claustrophobia, or other contraindications to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, PhD, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Aston Ambulatory Care Center, Allergy and Immunology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 patients were screened for eligibility between May 2012 and January 2016.
Pre-assignment Details: 46 of 73 participants were randomized. Of those not randomized, 27 did not meet inclusion criteria.
Period: First Intervention (24 Weeks)
Arm/Group | Memantine, Then Placebo | Placebo, Then Memantine
Started | 20 | 26
Completed | 14 | 23
Not Completed | 6 | 3
Period: Washout (4 Weeks)
Arm/Group | Memantine, Then Placebo | Placebo, Then Memantine
Started | 14 | 23
Completed | 14 | 22
Not Completed | 0 | 1
Period: Second Intervention (24 Weeks)
Arm/Group | Memantine, Then Placebo | Placebo, Then Memantine
Started | 14 | 22
Completed | 13 | 19
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Memantine, Then Placebo: Participants received Memantine 10 mg capsule twice/day for 24 weeks, then underwent a 4-week washout period, then received memantine-matched placebo capsule twice/day for 24 weeks.
  Memantine oral capsule was initiated at 5 mg/day at Week 0, then titrated to 5 mg twice/day at Week 2, then increased to 10 mg in the morning and 5 mg in the evening at Week 3, and then to 10 mg twice/day at Weeks 4-24. For the participants in the "Placebo, then Memantine" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
  Memantine-matched oral Placebo capsule was initiated at Week 0 and maintained Weeks 0-24 in a manner consistent with the active drug titration schedule. The number of placebo capsules matched the number of active drug capsules at each titration checkpoint. For the participants in the "Memantine, then Placebo" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
- Placebo, Then Memantine: Participants received Placebo capsule (matching Memantine 10 mg capsule) twice/day for 24 weeks. After a washout period of 4 weeks, they received Memantine 10 mg capsule twice a day for 24 weeks.
  Memantine oral capsule was initiated at 5 mg/day at Week 0, then titrated to 5 mg twice a day at Week 2, then increased to 10 mg in the morning and 5 mg in the evening at Week 3, and then to 10 mg twice a day (intervention dose) at Weeks 4-24. For the participants in the "Placebo, then Memantine" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
  Memantine-matched oral Placebo capsule was initiated at Week 0 and maintained Weeks 0-24 in a manner consistent with the active drug titration schedule. The number of placebo capsules matched the number of active drug capsules at each titration checkpoint. For the participants in the "Memantine, then Placebo" arm, the same titration schedule was maintained after the 4-week washout period (Week 28-52).
- Total: Total of all reporting groups
Arm/Group | Memantine, Then Placebo | Placebo, Then Memantine | Total
Number analyzed (Participants) | 20 | 26 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.10 (12.07) | 43.42 (12.72) | 43.28 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 18 | 27
Region of Enrollment [Number; unit: participants]
  United States | 20 | 26 | 46

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score
Description: Hopkins Verbal Learning Test-Revised (HVLT-R) is a word memory test that contains 12 nouns that are read to a participant for three consecutive trials. After each trial, a participant is asked to recall the words that were read to them. The number of words recalled on each trial is summed together to produce a total score. The total score (higher score means a better outcome) is converted to a standardized "T" score using normative data. The possible "T" score for each participant ranges from 20 to 80, with higher scores indicative of a better outcome.
Time Frame: Baseline and 24 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the analysis. Participants who dropped out during the washout period (between Weeks 24-28) did not receive the second intervention and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memantine: Participants who received Memantine 10 mg capsule twice per day in either the first or last 24 weeks of the study.
- Placebo: Participants who received placebo capsule (matching Memantine 10 mg) twice per day in either the first or last 24 weeks of the study.
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 42 | 40
units on a scale
  HVLT Total Score at Baseline | 39.40 (1.82) | 36.93 (1.72)
  HVLT Total Score at 24 weeks | 37.67 (1.61) | 38.37 (1.92)

ADVERSE EVENTS:
Time Frame: 24 weeks for each intervention.
Description: The safety population included all participants who received at least one dose of intervention.
Groups:
- Memantine: Participants who received Memantine 10 mg capsule twice per day for 24 weeks.
- Placebo: Participants who received Placebo capsule (matching Memantine 10 mg capsule) twice per day for 24 weeks.
Arm/Group | Memantine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 5/42 | 12/40
Other Adverse Events (participants affected / at risk) | 8/42 | 1/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=42) | Placebo (N=40)
Fournier's gangrene (Renal and urinary disorders) | 1 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
C. difficile (Infections and infestations) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Ear infection (Ear and labyrinth disorders) | 1 | 0
Gout flare (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypokalemia (Endocrine disorders) | 0 | 1
Lumbar spine injury (Injury, poisoning and procedural complications) | 0 | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Shingles (Infections and infestations) | 0 | 1
Lupus flare (Skin and subcutaneous tissue disorders) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 2
Vulvar squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=42) | Placebo (N=40)
Abnormal stool color (Gastrointestinal disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Elevated blood pressure (Vascular disorders) | 1 | 0
Low blood pressure (Vascular disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pregnancy (Reproductive system and breast disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Elevated blood glucose (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No